CLINICAL TRIAL: NCT07114679
Title: Molecular Breast Imaging (MBI)-Guided Biopsy Pilot SBIR
Brief Title: Molecular Breast Imaging (MBI)-Guided Biopsy
Acronym: MBI-GB-Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Breast Corp. (Industry)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MBI_Biopsy_Pilot_SBIR
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Detection; Breast Neoplasm; Molecular Imaging; Biopsy; Dense Breasts
Keywords: screening; crossover; single-group; pilot; biopsy; randomized assignment; dense breasts; MBI; molecular imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Every participant (dense breast woman) will receive both screening DBT and screening MBI (crossover). If biopsy is required, participant will be randomly assigned to either DBT-guided or MBI-guided biopsy.
Masking Description: After MBI-guided biopsy samples are placed sequentially in a Petri dish, an MBI image of the samples is taken. This image will be compared to the pathology report for concordance. The Outcomes Assessor will be blinded to patient ID and medical records. Similarly, the pathology report and screening DBT images will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Breast screening (Active Comparator): Screening DBT and screening MBI are compared in women with dense breasts. Then, DBT-guided biopsy and MBI-guided biopsy are compared.
  Interventions: Device: Molecular Breast Imaging; Device: MBI-guided biopsy

INTERVENTIONS:
Device: Molecular Breast Imaging — MBI is a molecular imaging (nuclear medicine) technique using a low dose i.v. radiopharmaceutical injection and solid-state gamma cameras to image the breast, where cancer mitochondria avidly take up the radiopharmaceutical.
  Other Names: MBI
Device: MBI-guided biopsy — Two stereotactic MBI views of the breast produce a precise 3D location for each lesion targeted for biopsy. A vacuum-assisted core biopsy needle is guided to the lesion position.

SUMMARY:
The goal of this pilot clinical trial is to demonstrate supplemental screening MBI (molecular breast imaging) in women with dense breasts. The main questions it aims to answer are:

* Does screening MBI find more cancer than screening DBT (3D mammography, digital breast tomosynthesis?
* Does screening MBI result in more call-backs for biopsy than DBT?
* How well does MBI-guided biopsy conform with pathology reports?

Researchers will compare screening MBI to screening DBT to see if MBI is more sensitive to detecting cancer in women with dense breasts.

Participants will

* Receive both screening DBT and screening MBI
* Receive either DBT-guided or MBI-guided biopsy (randomly assigned), if required by the screening images

DETAILED DESCRIPTION:
This is a pilot single-group crossover screening clinical trial comparing screening MBI (molecular breast imaging) to screening DBT (3D mammography, digital breast tomosynthesis. Women who have recently completed their annual screening DBT will be assessed for breast density. If they have BI-RADS density C or D (dense breasts), they are eligible for this study. After consent, participants will receive a supplemental screening MBI (crossover from DBT). Both screenings will be read while blinded to knowledge of the other. After independent reporting, a Conciliation Conference will compare the two, and a consensus report will be prepared.

If biopsy is required on the consensus basis of both image sets, then the participant will be randomly assigned to DBT-guided or MBI-guided biopsy. If only one modality has visible lesions that require biopsy, then that modality will be assigned.

The primary outcome measure is Cancer Detection Rate. Secondary outcome measures include Biopsy Callback Rate, Concordance Rate between MBI biopsy sample images and pathology, Time Duration of Biopsy, and Accuracy of Lesion Targeting.

ELIGIBILITY:
Inclusion Criteria:

* dense breasts (BI-RADS C or D) on screening DBT

Exclusion Criteria:

* pregnancy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2027-06 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate | less than one day
  The number of cancers found by a particular modality compared to the number of women with dense breasts screened by that modality.

SECONDARY OUTCOMES:
Concordance Rate | less than a day
  MBI-guided biopsies include an MBI image of the biopsy tissue samples in a Petri dish. Comparison of that image with the pathology report yields concordance.
Biopsy Call-Back Rate | less than a day
  The percentage of women with dense breasts screened by a particular modality who have a suspicious lesion on their screening and they require biopsy.
Duration of Biopsy | less than a day
  The amount of time that the modality-guided biopsy took to complete.

CONTACTS AND LOCATIONS:
Overall Officials: James W Hugg, PhD, Principal Investigator — Smart Breast Corp.
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We will reconsider at the end of data acquisition.